CLINICAL TRIAL: NCT06333613
Title: Evaluation of Acuvue Oasys 1-Day Contact Lenses in New Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6565
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Test Lens (Experimental): Eligible subjects will be fitted bilaterally with the TEST lens for approximately 2 weeks of wear (two 1-week wear periods).
  Interventions: Device: ACUVUE OASYS® 1-DAY with HydraLuxe™ TECHNOLOGY (AO1D)

INTERVENTIONS:
Device: ACUVUE OASYS® 1-DAY with HydraLuxe™ TECHNOLOGY (AO1D) — Test Lens

SUMMARY:
This is a multi-site, bilateral, dispensing, non-randomized, uncontrolled, unmasked, single arm study to evaluate visual acuity in neophytes.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

The subject must:

1. Read, understand, and sign the Statement of Informed Consent and receive a fully executed copy of the form (For subjects aged 18 and older)
2. Read (or be read to) and sign the Children's Assent (Information and Assent Form) and receive a fully executed copy of the form. (For subjects aged 13 to 17)
3. Have parents or legal guardians who must read, understand, and sign the Statement of Informed Consent (Parental Permission Form and Authorization to Use and Disclose Medical Information). (For subjects aged 13 to 17)
4. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
5. Be between 13 and 39 (inclusive) years of age at the time of screening.
6. By self-report, having never worn any type of contact lenses and never attempted to insert contact lenses.
7. Have a pair of prescription glasses on hand that corrects distance vision, if determined to be required by the investigator.
8. The magnitude of the cylindrical component of the subject's vertex-corrected distance refraction must be ≤ 0.75 DC in each eye.
9. Subject must have a vertex corrected distance sphero-cylindrical refraction in the range such that appropriate spherical lens powers are available for correction in both eyes. The spherical lens powers available in this study are:

   a. -1.00 to -6.00 (in 0.25D steps)
10. Best corrected monocular distance visual acuity must be 20/20-3 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The subject must not:

1. Be currently pregnant or lactating.
2. Be currently using any ocular medications or have any ocular infection of any type.
3. By self-report, have any ocular or systemic disease, allergies, or infection, or use medications that the investigator believes might contraindicate or interfere with contact lens wear, or otherwise compromise the study endpoints. See section 9.1 for additional details regarding systemic medications.
4. Have previously participated in a contact lens, contact lens package, or lens care related clinical trial.
5. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild, or sibling of the employee or their spouse) of the clinical site.
6. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings or other corneal, eyelid, or ocular disease or abnormalities that the investigator believes might contraindicate contact lens wear or may otherwise compromise study endpoints (including significant blepharitis, entropion, ectropion, ptosis, chalazia, recurrent styes, pterygium, significant dry eye disease, history of recurrent corneal erosions, aphakia, corneal distortion, herpetic keratitis).
7. Have a history of strabismus or amblyopia.
8. Have fluctuations in vision due to clinically significant dry eye or other ocular or systemic conditions.
9. Have had or have planned (within the study period) any ocular or intraocular surgery or procedures (e.g., PRK, LASIK, IPL, blepharoplasty, etc.)

Ages: 13 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (5):
- United States (5):
  - Scripps Poway Eyecare & Optometry, San Diego, California
  - Omega Vision Center, Longwood, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Procare Vision Centers, Granville, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 36 subjects were enrolled in this study. Of those enrolled, 34 subjects were dispensed the study lens, while 1 subject withdrew consent before lens dispensing and 1 subject failed to meet all eligibility criteria. Of those dispensed, 33 subjects completed the study while 1 subject was discontinued.
Groups:
- Test (Senofilcon A C3): All eligible subjects were dispensed the study lens.
Period: Overall Study
Arm/Group | Test (Senofilcon A C3)
Started | 34
Completed | 33
Not Completed | 1
Not completed — Doesn't Like Wearing Contacts | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.1 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 1
  White | 28
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Incidence (Percentage) of Eyes With Grade 3 or 4 Slit Lamp Findings Related to the Study Lenses
Description: Slit Lamp Findings (SLFs) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). SLF assessment was performed on each subject eye at different study visits (Baseline, unscheduled visits, 1-week follow-up, 2-Week Follow-up, and Final Evaluation). The percentage of eyes with SLF of grade 3 or grade 4 was reported.
Time Frame: Up to 2-Week Follow-up
Population: All dispensed subjects regardless of subsequent withdrawal from study or deviation from protocol.
Measure: Number; unit: Percentage
Units Other Than Participants: Eyes
Groups:
- Test (Senofilcon A C3): All subjects that were dispensed the Test lens.
Arm/Group | Test (Senofilcon A C3)
Number analyzed (Participants) | 34
Number analyzed (Eyes) | 68
Percentage | 0

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 2-weeks per subject.
Description: All subjects dispensed the study lens.
Groups:
- Test (Senofilcon A C3): All subjects dispensed the study lens.
Arm/Group | Test (Senofilcon A C3)
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT06333613/Prot_SAP_000.pdf